CLINICAL TRIAL: NCT03799913
Title: A Clinical Trial of MESO-CAR T Cells Therapy for Relapsed and Refractory Ovarian Cancer
Brief Title: MESO-CAR T Cells Therapy for Relapsed and Refractory Ovarian Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Hrain Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhigang Zhang, Dr, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESO
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Cancer
Keywords: CAR-T; MESO; Ovarian Cancer; Relapsed and Refractory
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-MESO CAR-T cells (Experimental): Administration with anti-MESO CAR-T cells in the MESO-positive ovarian cancer patients
  Interventions: Biological: anti-MESO CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-MESO CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-MESO CARs
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 300mg/m2/d

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-MESO antigen receptors (CARs) T cell therapy for relapsed and refractory ovarian cancer.

DETAILED DESCRIPTION:
Primary Objectives

1.To determine the feasibility ad safety of anti-MESO CAR-T cells in treating patients with MESO-positive ovarian cancer.

Secondary Objectives

1. To access the efficacy of anti-MESO CAR-T cells in patients with ovarian cancer.
2. To determine in vivo dynamics and persistency of anti- MESO CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 Years Old, female;
2. Expected survival > 12 weeks;
3. Clinical performance status of ECOG score 0-2;
4. Patients who have previously been treated with second- line or more lines of standard treatment are not effective (No remission or recurrence after remission);
5. At least one measurable tumor foci according to RECIST standard 1.1 ;
6. Positive Mesothelin expression in tumor tissues;
7. Creatinine ≤ 1.5×ULN;
8. ALT and AST ≤ 3×ULN;
9. Total bilirubin ≤ 2×ULN;
10. Hemoglobin≥90g/L;
11. Absolute counting of neutrophils≥1000uL ;
12. Absolute counting of lymphocytes>0.7×10^9/L;
13. Counting of Platelet≥75000/uL;
14. The venous access required for collection can be established without contraindications for leukocyte collection;
15. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. Accompanied by other uncontrolled malignant tumors;
2. Active hepatitis B, hepatitis C, syphilis, HIV infection;
3. Suffering severe cardiovascular or respiratory disease;
4. Any other diseases could affect the outcome of this trial;
5. Any affairs could affect the safety of the subjects or outcome of this trial;
6. Pregnant or lactating women, or patients who plan to be pregnancy during or after treatment;
7. There are active or uncontrollable infections (except simple urinary tract infections or upper respiratory tract infections) that require systemic therapy 14 days or 14 days prior to assignment;
8. Patients who are accounted by researchers to be not appropriate for this test;
9. Received CAR-T treatment or other gene therapies before assignment;
10. Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 1 years post infusion

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 12 months post infusion
Progress Free Survival (PFS) after administration | 12 months post infusion
Duration of CAR-positive T cells in circulation | 12 months post infusion
Detection of PD1 antibody in serum | 12 months post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Zhou, M.D., Study Chair — Zhejiang University
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No